CLINICAL TRIAL: NCT04065139
Title: Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) in Gastric Carcinomatosis. Phase II Randomized Study - PIPAC EstoK 01
Brief Title: Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) in Gastric Carcinomatosis. Phase II Randomized Study
Acronym: PIPAC EstoK 01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P160951J; 2018-004755-20 (EudraCT Number)
Record Dates: First submitted 2019-08-21; First posted 2019-08-22 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Gastric Adenocarcinoma; Cancer Metastatic; Chemotherapy Effect
Keywords: pressurized intraperitoneal aerosol chemotherapy (PIPAC); gastric adenocarcinoma; metastasis
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Active Comparator)
  Interventions: Drug: Standard chemotherapy
- Experimental Arm : PIPAC (Experimental)
  Interventions: Drug: Pressurized intraperitoneal aerosol chemotherapy (PIPAC)

INTERVENTIONS:
Drug: Pressurized intraperitoneal aerosol chemotherapy (PIPAC) — After insufflation of a 12 mmHg of capnoperitoneum at 37°C, two balloons safety trocars (10 and 12mm) are inserted into the abdominal wall. Injection of Doxorubicin (2.1 mg/m2 in 50 ml NaCl 0.9%) and Cisplatin (10.5 mg/m2 body surface in 150 ml NaCl 0.9%) with a flow rate of 0.7ml/s, the therapeutic capnoperitoneum is maintained for 30 min at body temperature.
  Arms: Experimental Arm : PIPAC
Drug: Standard chemotherapy — Patient will receive standard poly chemotherapy proposed by the oncologist or any new standard validated during the study, until progression or toxicity.
  Arms: Control Arm

SUMMARY:
Peritoneal metastasis is a common pattern in advanced gastric cancer leading to a terminal condition in a very short time. Whatever recent progress regarding systemic chemotherapy using multi drugs association median survival is limited to 6 months with altered quality of life (QoL) after 4 months for all patients. We postulated that a new innovative health technology for delivering intraperitoneal pressurized aerosol of chemotherapy (Doxorubicin and Cisplatin) during laparoscopy can transform that situation offering to double the survival with QoL preservation. Interestingly, PIPAC procedure is made to be applied repeatedly, every 4 to 6 weeks. This therapeutic strategy allows to improved Intra Peritoneal (IP) drugs impregnation and maintained Intra-Veinous (IV) chemotherapy meanwhile. The primary objective of this study is to evaluate and compare 24-month progression free-survival in patients with peritoneal carcinomatosis of gastric cancer treated either with IV chemotherapy and Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) or with IV chemotherapy alone, with preservation of quality of life.

ELIGIBILITY:
Inclusion Criteria:

* 18 < age ≤ 75 years
* Performance status (WHO) < 2
* White blood cells > 3.500 /mm3; neutrophils > 1.500 /mm3; platelets > 100.000 /mm3
* Creatinemia < 1.5 x Normal, Normal ASAT, ALAT and Serum total bilirubin, Normal ionic balance (potassium, calcium, magnesium and phosphorus
* An acceptable nutritional condition with Body Mass Index (BMI) > 18.5 kg/m2, Albumin > 30 g/l, pre-albumin > 110 mg/l
* Effective contraception for patients of childbearing age
* Written consent obtained prior any act of the research
* Patient with social insurance
* Patient having synchronous or metachronous peritoneal metastasis or ovarian metastasis of a gastric adenocarcinoma cancer, including adenocarcinoma with independent cells (ADCI) or linitis
* Patients with or without primary gastric tumor could be included
* Peritoneal Cancer Index (PCI) > 8

Exclusion Criteria:

* Weight loss > 20% of total body weight before disease
* Presence of uncontrolled comorbidities including severe chronic disease or organ insufficiency
* Contraindication to any drug contained in the chemotherapy regimen, according to summary of product characteristic's
* Having any form of previous intra-abdominal chemotherapy or intra-abdominal antibody therapy
* Patients with history of allergic reactions to platinum compounds or doxorubicin
* Complete deficiency of the enzyme dihydropyrimidine dehydrogenase.
* Patients are not allowed to undergo any cancer-specific treatment during the trial.
* Secondary debulking surgery is not allowed during PIPAC treatment
* Pregnancy or breastfeeding
* Patient under guardianship
* Other systemic metastases (liver, lung, bone, brain) or lombo-aortic lymph node involvement
* Pleural effusion requiring evacuation for respiratory failure
* Small bowel occlusion with no possible food intake
* Ascites > 3 liters
* HER2 +++ tumor

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2024-03-02 (Actual); Study Completion 2024-03-02 (Actual)

PRIMARY OUTCOMES:
Progression Free survival | 24 months
  24-month progression free-survival, defined as time from randomization to any clinical (ascites, abdominal pain, weight loss > 10% of total body weight) and/or morphological signs (systemic metastases, ascites, progression with RECIST criteria) of recurrence (local or systemic) or death.

SECONDARY OUTCOMES:
Postoperative pain H6 | 6 hours after end of surgery
  Postoperative pain with a numeric rating scale from 0 to 10 (0 being no pain and 10 the worst possible pain)
Postoperative pain H12 | 12 hours after end of surgery
  Postoperative pain with a numeric rating scale from 0 to 10 (0 being no pain and 10 the worst possible pain)
Postoperative pain H18 | 18 hours after end of surgery
  Postoperative pain with a numeric rating scale from 0 to 10 (0 being no pain and 10 the worst possible pain)
Postoperative pain H24 | 24 hours after end of surgery
  Postoperative pain with a numeric rating scale from 0 to 10 (0 being no pain and 10 the worst possible pain)
Postoperative pain H30 | 30 hours after end of surgery
  Postoperative pain with a numeric rating scale from 0 to 10 (0 being no pain and 10 the worst possible pain)
Postoperative pain H36 | 36 hours after end of surgery
  Postoperative pain with a numeric rating scale from 0 to 10 (0 being no pain and 10 the worst possible pain)
Postoperative pain H42 | 42 hours after end of surgery
  Postoperative pain with a numeric rating scale from 0 to 10 (0 being no pain and 10 the worst possible pain)
Postoperative pain H48 | 48 hours after end of surgery
  Postoperative pain with a numeric rating scale from 0 to 10 (0 being no pain and 10 the worst possible pain)
Overall survival | 24 months
  Progression Free survival
Secondary resectability rate | 24 months
  Secondary resectability rate after the treatment
Quality of life | monthly until death or 24 months
  Quality of life evaluated monthly by the patient with the EORTC QLQ-STO22 questionnaire
Quality of health status | monthly until death or 24 months
  Quality of health status evaluated monthly by the patient with the EQ-5D-5L questionnaire
Toxicity | 60 days
  Rate of treatment-related toxicity at 60 days of each PIPAC procedure
PIPAC success | 24 hours
  Rate of successful PIPAC procedures
Morbidity Clavien-Dindo | 60 days
  Morbidity will be evaluated on post-operative day 60 by the Clavien-Dindo classification (I to V)
Morbidity Complication Index | 60 days
  Morbidity will be evaluated by the Comprehensive Complication Index, ranging from 0 to 100 (https://www.assessurgery.com/about_cci-calculator)
Discontinuation | 24 months
  The time of discontinuation defined as the time from randomization to therapy change or dose reduction because of progression of disease or intolerance or adverse effects or patient refusal or death.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Universitaire Claude Huriez, Lille, France

IPD SHARING:
Plan to Share IPD: Undecided